CLINICAL TRIAL: NCT00109226
Title: A Phase II, Multicenter, Double-Blind, Randomized, Active-Controlled Clinical Trial to Evaluate the Efficacy and Safety of rhuMAb VEGF (Bevacizumab), a Recombinant Humanized Monoclonal Antibody to Vascular Endothelial Growth Factor, in Combination With 5-Fluorouracil and Leucovorin Chemotherapy in Subjects With Metastatic Colorectal Cancer Who Are Not Optimal Candidates for First Line CPT-11
Brief Title: A Study to Evaluate Avastin in Combination With Chemotherapy in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: AVF2192g; NCT00012272 (obsolete NCT alias)
Record Dates: First submitted 2005-04-26; First posted 2005-04-26 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Bevacizumab

INTERVENTIONS:
Drug: Avastin (Bevacizumab)

SUMMARY:
This Phase II, multicenter, double-blind, randomized, active-controlled trial is designed to evaluate the efficacy and safety of rhuMAb VEGF (Avastin) when administered at a dose of 5 mg/kg every 2 weeks in combination with 5 FU (fluorouracil)/leucovorin versus 5 FU/leucovorin alone in subjects with previously untreated metastatic colorectal cancer who are not optimal candidates to receive first-line CPT-11 (irinotecan). A total of 48 doses of rhuMAb VEGF may be administered during this study (maximum of 96 weeks of therapy).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age >=18 years
* Use of an effective means of contraception in women of childbearing potential
* Histologically confirmed (resected or biopsied primary tumor) colorectal carcinoma with evidence of metastases (i.e., by radiographic imaging or biopsy)
* Ability to tolerate CT contrast dye.
* Bi-dimensionally measurable disease (minimum of two lesions)
* Life expectancy of >3 months
* Willingness and capability to be accessible for follow-up until death
* In addition, subjects must meet at least one of the following criteria to be eligible for study entry: *Age >=65 years; *ECOG performance status of 1 or 2; *Albumin <=3.5 g/dL; *Prior radiotherapy to the abdomen or pelvis; and, *in the opinion of the treating physician, not be an optimal candidate for first-line CPT-11

Exclusion Criteria:

* Prior administration of chemotherapy other than adjuvant fluoropyrimidines in combination with leucovorin and/or levamisole
* Administration of adjuvant fluoropyrimidines in combination with leucovorin and/or levamisole completed <=12 months prior to Day 0
* Administration of fluoropyrimidines as a radiosensitizer during pelvic radiotherapy for rectal cancer completed <=12 months prior to Day 0
* Prior radiotherapy to a measurable, metastatic lesion(s) to be used to measure response
* Radiotherapy within 14 days prior to Day 0
* Prior administration of biotherapy for colorectal cancer
* Evidence of clinically detectable ascites prior to Day 0
* Other invasive malignancies within 5 years of Day 0 (other than basal cell carcinoma of the skin)
* History or evidence upon physical examination of CNS disease (e.g., primary brain tumor, seizures not controlled with standard medical therapy, or any brain metastases)
* Serious, nonhealing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure within 28 days prior to Day 0, or open biopsy, significant traumatic injury, or anticipation of need for major surgical procedure during the course of the study; fine needle aspirations within 7 days prior to Day 0
* Current or recent (within the 10 days prior to Day 0) use of oral or parenteral anticoagulants (except as required to maintain patency of preexisting, permanent indwelling IV catheters) or thrombolytic agent
* Chronic, daily treatment with aspirin (>325 mg/day) or nonsteroidal anti-inflammatory medications (of the kind known to inhibit platelet function)
* Pregnancy (positive pregnancy test) or lactation
* Proteinuria at baseline or clinically significant impairment of renal function
* Current or recent (within 28 days prior to Day 0) participation in another experimental drug study
* Active infection requiring parenteral antibiotics on Day 0
* Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, myocardial infarction, unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix H), serious cardiac arrhythmia requiring medication, or Grade II or greater peripheral vascular disease within 1 year prior to Day 0
* ECOG performance status of >2
* Screening clinical laboratory values: *ANC of <=1500/uL; *Platelet count of <=75,000/uL; *International normalized ratio (INR) of >=1.5; *Total bilirubin of >2.0 mg/dL; *AST or ALT of >=5 times the upper limit of normal for subjects with documented liver metastases; >2.5 times the upper limit of normal for subjects without evidence of liver metastases; *Serum creatinine of >2.0 mg/dL; *Hemoglobin of <9 gm/dL (may be transfused to maintain or exceed this level); *Proteinuria (24-hour urine collection demonstrated >=500 mg of protein/24 hr)
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications
* Inability to comply with the study visit and follow-up schedule or procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Study Completion 2003-09 (Actual)

REFERENCES:
- [Result] Scappaticci FA, Skillings JR, Holden SN, Gerber HP, Miller K, Kabbinavar F, Bergsland E, Ngai J, Holmgren E, Wang J, Hurwitz H. Arterial thromboembolic events in patients with metastatic carcinoma treated with chemotherapy and bevacizumab. J Natl Cancer Inst. 2007 Aug 15;99(16):1232-9. doi: 10.1093/jnci/djm086. Epub 2007 Aug 8. PMID 17686822
- [Result] Kabbinavar FF, Wallace JF, Holmgren E, Yi J, Cella D, Yost KJ, Hurwitz HI. Health-related quality of life impact of bevacizumab when combined with irinotecan, 5-fluorouracil, and leucovorin or 5-fluorouracil and leucovorin for metastatic colorectal cancer. Oncologist. 2008 Sep;13(9):1021-9. doi: 10.1634/theoncologist.2008-0003. Epub 2008 Sep 5. PMID 18776057
- [Result] Kabbinavar FF, Hurwitz HI, Yi J, Sarkar S, Rosen O. Addition of bevacizumab to fluorouracil-based first-line treatment of metastatic colorectal cancer: pooled analysis of cohorts of older patients from two randomized clinical trials. J Clin Oncol. 2009 Jan 10;27(2):199-205. doi: 10.1200/JCO.2008.17.7931. Epub 2008 Dec 8. PMID 19064978